CLINICAL TRIAL: NCT06791252
Title: The Effect of Genital Hygiene Education Given to Pregnant Women Diagnosed with Urinary Tract Infection on Genital Hygiene Behavior and Self-Care Agency
Brief Title: Genital Hygiene Education and Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, ESRA GUNEY, PhD, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/2261
Record Dates: First submitted 2025-01-16; First posted 2025-01-24 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2022-02

CONDITIONS: Genital Hygiene Behaviors; Self-Care Ability
Keywords: Midwife; pregnant; hygiene; self-care; urinary tract infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: randomized controlled trial conducted with experimental and control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group receiving genital hygiene education (Experimental): Pregnant women in the experimental group were given genital hygiene training in 4 sessions.
  Interventions: Behavioral: genital hygiene education
- Control Group (No Intervention): No intervention was applied to the control group other than the application of data collection tools simultaneously with the pregnant women in the experimental group (pre-test: 1st session/1st day - post-test: 2nd session/30th day).

INTERVENTIONS:
Behavioral: genital hygiene education — The pregnant women in the experimental group were given genital hygiene training individually and in their own homes by the researcher. During the training, the privacy of the client was observed and the researcher and the pregnant women were left alone in the room where the training would be given. Care was taken to ensure that the environment was quiet and calm while the training was given. It was preferred that the pregnant women be in the most comfortable position during the training.
  The training was completed by explaining each topic in the training booklet in an average of 20-25 minutes.
  Genital hygiene training content:
  Session 1 (Day 1): After the introduction phase, information was given about the method to be followed in the study to the pregnant women who agreed to participate in the study. Then, the "Minimum Informed Consent Form" was given to these women, and the pregnant women who approved the form after reading it were included in the study. Pre-test data were collecte
  Arms: Group receiving genital hygiene education

SUMMARY:
Genital hygiene behaviors are of great importance in preventing urinary tract infections, especially during pregnancy. The study was conducted to determine the effect of genital hygiene education given to pregnant women diagnosed with urinary tract infections on genital hygiene behavior and self-care ability. The hypotheses of this study were determined as follows:

H1a: Genital hygiene education affects genital hygiene behavior in pregnant women.

H1b: Genital hygiene education affects self-care ability in pregnant women.

DETAILED DESCRIPTION:
Genital hygiene behaviors are of great importance in preventing urinary tract infections, especially during pregnancy. The study was conducted to determine the effect of genital hygiene education given to pregnant women diagnosed with urinary tract infection on genital hygiene behavior and self-care ability. The study was conducted in the gynecology and obstetrics clinics of a hospital in eastern Turkey between September 2021 and February 2022. Personal Information Form, Genital Hygiene Behaviors Scale and Self-Care Ability Scale were used to collect data. In the power analysis, the sample size was calculated as 80 pregnant women in each group (80 experimental, 80 control). Pregnant women in the experimental group received genital hygiene education in 4 sessions, while no intervention was applied to the control group. Descriptive statistical analyses and t-test in dependent-independent groups were used in the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who were literate, - Who had completed their pharmacological treatment (antibiotic treatment) for UTI according to medical records were included in the sample

Exclusion Criteria:

* - Those who had previously received training to increase genital hygiene behavior,
* Those who had a risky pregnancy,
* Those who were diagnosed with any health problems related to the pregnant woman and the fetus were not included in the study

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women
Enrollment: 80 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
genital hygiene behavior | 30 days
  Considering that behaviors regarding genital hygiene are established from an early age, it is important to objectively determine risky behaviors in young women who are not yet sexually active in order to take precautions for improving genital hygiene.In this way, many negative outcomes that may occur during the fertile period and are directly related to genital infections, such as infertility, abortion, and the threat of premature birth,can be prevented.On the other hand, it would be useful to use an objective, valid, and reliable measurement tool in determining the relationship between genital hygiene behaviors in women and situations such as the threat of premature birth, premature rupture of membranes, and postpartum infection.The primary outcome of this study is to determine the genital hygiene behaviors of the hygiene education given to women who have previously had urinary tract infections.For this purpose, the General Hygiene Habit and Abnormal Finding Awareness scale was used.

SECONDARY OUTCOMES:
Self-Care Ability | 30 days
  Self-care is the activities initiated and carried out by an individual to protect, maintain and improve their life, health and well-being. According to Orem, self-care needs are divided into three groups: universal, developmental and self-care needs in deviations from health. Universal needs are special care behaviors that occur at different developmental levels of the individual, such as infancy, childhood and pregnancy. Pregnancy is also a developmental condition and is a subject that should be examined separately due to its importance. During pregnancy, a woman may need help if her health deteriorates and she cannot meet her care needs. It is important to use an objective, valid and reliable measurement tool in determining the relationship between the self-care of pregnant women and conditions such as urinary system infections. In this study, self-care power was determined as a secondary outcome and the self-care power scale was used to determine the effect of hygiene training give

CONTACTS AND LOCATIONS:
Locations (1):
- Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Research results will be shared

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29402148/